CLINICAL TRIAL: NCT01853501
Title: Effects of Adipose Derived Stem Cell Therapy in Women With Premature Ovarian Failure
Brief Title: Effects of ADSC Therapy in Women With POF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Nanjing University (Other)
Responsible Party: Principal Investigator, Li-jun Ding, lecturer, Nanjing University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 973 Project No. 2010CB945 104
Record Dates: First submitted 2013-05-07; First posted 2013-05-15 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2013-11

CONDITIONS: Premature Ovarian Failure
Keywords: POF
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- POF,treatment,ADSC (Experimental): Fat from POF patients undergo Autologous fat grafting operation were separated, from which Adipose Derived Stem Cell were then purified and injected into the both ovaries of patients.
  Interventions: Procedure: Autologous fat grafting

INTERVENTIONS:
Procedure: Autologous fat grafting — ADSC ovary injection

SUMMARY:
The purpose of this study is to determine whether Adipose Derived Stem Cells are effective in the treatment of Premature Ovarian Failure (POF). Stem cell transplantation has been reported to rescue ovarian function in a pre-clinical mouse model of chemotherapy-induced POF; however, maintaining the survival of transplanted cells in human ovarian tissues to enable the POF patients regain ovary function over the long-term and achieving a successful pregnancy remain a troublesome issue. In this study the investigators are aiming to determine whether the CD29+/CD44+ human Adipose Derived Stem Cells could later enable ovaries produce mature oocytes.

DETAILED DESCRIPTION:
The purpose of this study was to explore the therapeutic potency of the adipose derived stem cells (ADSC) transplantation for premature ovarian failure (POF) women underwent Autologous fat transplantation. The serum of each patient were kept and sent for laboratory test before the surgery. 100ml fat was harvested from the abdomen of POF patient using abdominal fat abortion. And ADSC were isolated and cultured in vitro using autologous serum. The biomarkers of ADSC, CD29 and CD44, were detected in the ADSC cultures using Flow cytometry detection. The ADSC were then transplanted directly into bilateral ovaries when cells reach a density of 5-10×106. The clinical conditions of patients were examined at 1, 2, 4 and 8 weeks after the transplantation. Ovarian functions were evaluated by follicle diameter and sexual hormone levels. The follicle number was counted and radiology data were kept for future analysis. To ensure high rate of pregnancy, intercourse under medical guidance may be suggested and hormone replacement treatment may be taken to help the patients conceive.

Main Outcome Measure(s): Serum FSH,LH,E2 levels, recurrence of Menstruation, Antral follicle diameter,and pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Premature Ovarian Failure
* Patients show no response to drug treatment
* Willing to receive follow up
* Willing to conceive a baby
* Age between 20 to 39

Exclusion Criteria:

* Patients with few abdominal fat
* Patients with chromosome abnormalities
* Patients with congenital ovarian malformations
* Patients with severe endometriosis
* Patients with thyroid dysfunction
* Patients with pregnancy contraindications
* Patients with hormone replacement therapy contraindications
* Patients with liposuction contraindications
* Past history of ovarian tumors or after radiotherapy
* Can not take the follow-up, or want to take other treatment during the follow-up period
* Patients with immune system diseases

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Estimated)
Dates: Start 2012-09; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Antral follicle diameter | within the first 30 weeks (plus or minus 10 weeks) after surgery
  Antral follicle diameter were record using transvaginal ultrasound scan.

CONTACTS AND LOCATIONS:
Overall Officials: Yali Hu, Ph.D., Principal Investigator — The Affiliated Drum Tower Hospital of Nanjing University
Locations (1):
- The Affiliated Drum Tower Hospital of Nanjing University, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Silber SJ. Ovary cryopreservation and transplantation for fertility preservation. Mol Hum Reprod. 2012 Feb;18(2):59-67. doi: 10.1093/molehr/gar082. Epub 2011 Dec 28. PMID 22205727
- [Background] Lin G, Wang G, Banie L, Ning H, Shindel AW, Fandel TM, Lue TF, Lin CS. Treatment of stress urinary incontinence with adipose tissue-derived stem cells. Cytotherapy. 2010;12(1):88-95. doi: 10.3109/14653240903350265. PMID 19878076
- [Background] Cho WK, Lee JW, Chung NG, Jung MH, Cho B, Suh BK, Kim HK. Primary ovarian dysfunction after hematopoietic stem cell transplantation during childhood: busulfan-based conditioning is a major concern. J Pediatr Endocrinol Metab. 2011;24(11-12):1031-5. doi: 10.1515/jpem.2011.339. PMID 22308860
- [Background] Feng W, Cui Y, Zhan H, Shi M, Cui W, Guo K, Li Q, Song C, Zhang Y, Mori T, Gershwin ME, Abraham NG, Ikehara S. Prevention of premature ovarian failure and osteoporosis induced by irradiation using allogeneic ovarian/bone marrow transplantation. Transplantation. 2010 Feb 27;89(4):395-401. doi: 10.1097/TP.0b013e3181ca86bb. PMID 20177340
- [Result] Takehara Y, Yabuuchi A, Ezoe K, Kuroda T, Yamadera R, Sano C, Murata N, Aida T, Nakama K, Aono F, Aoyama N, Kato K, Kato O. The restorative effects of adipose-derived mesenchymal stem cells on damaged ovarian function. Lab Invest. 2013 Feb;93(2):181-93. doi: 10.1038/labinvest.2012.167. Epub 2012 Nov 19. PMID 23212100
- See also: IVF center website — http://www.ivf-gl.com/